CLINICAL TRIAL: NCT07241611
Title: Role of Cervical Fascia Flap in Decreasing the Incidence of Pharyngocutaneous Fistula After Total Laryngectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MS.24.08.2855
Record Dates: First submitted 2025-11-14; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Malignant Tumor of the Larynx
MeSH Terms: conditions — Laryngeal Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cervical fascia flap group (Active Comparator)
  Interventions: Procedure: Total laryngectomy
- conventional repair group (Active Comparator)
  Interventions: Procedure: Total laryngectomy

INTERVENTIONS:
Procedure: Total laryngectomy — pharyngeal repair after total larygectomy

SUMMARY:
This study was conducted to evaluate the potential role of using the cervical fascia flap over the pharyngeal closure line to enhance healing and subsequently to decrease the incidence of pharyngocutaneous fistula after total laryngectomy.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive patients who will undergo total laryngectomy for advanced laryngeal carcinoma in the study duration.

Exclusion Criteria:

* Presence of extra-laryngeal extension.
* Patients undergoing partial pharyngectomy.
* Previous neck irradiation.
* Previous neck surgery.
* Patients' refusal to participate in the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
incidence of pharyngocutaneous fistula after total laryngectomy | Four weeks

SECONDARY OUTCOMES:
subjective assessment of the swallowing function after surgery | three months
  swallowing was evaluated subjectively by applying the Eating Assessment Tool (EAT-10) questionnaire
objective assessment of the swallowing function after surgery | Three months
  swallowing was evaluated objectively by functional endoscopic evaluation of swallowing (FEES)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Mansoura University, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zorlu ME, Kertmen C, Aysel A, Yilmaz F, Dalgic A, Muderris T. Use of Cervical Fascia to Prevent Pharyngocutaneus Fistula After Total Laryngectomy. Laryngoscope. 2024 Dec;134(12):4964-4970. doi: 10.1002/lary.31606. Epub 2024 Jun 28. PMID 38940495
- [Background] Wang M, Xun Y, Wang K, Lu L, Yu A, Guan B, Yu C. Risk factors of pharyngocutaneous fistula after total laryngectomy: a systematic review and meta-analysis. Eur Arch Otorhinolaryngol. 2020 Feb;277(2):585-599. doi: 10.1007/s00405-019-05718-9. Epub 2019 Nov 11. PMID 31712878
- [Background] Eid AM, Ebada HA, El-Fattah AMA, Tawfik A. Platelet-rich fibrin: an autologous biomaterial for healing assistance of pharyngeal repair in total laryngectomy. Eur Arch Otorhinolaryngol. 2021 Feb;278(2):463-470. doi: 10.1007/s00405-020-06404-x. Epub 2020 Oct 3. PMID 33009930
- [Background] Park J, Chang C, Kwon D. Use of fibrin adhesive for preventing pharyngocutaneous fistula in total laryngectomy. Am J Otolaryngol. 2020 Nov-Dec;41(6):102674. doi: 10.1016/j.amjoto.2020.102674. Epub 2020 Aug 13. PMID 32836041